CLINICAL TRIAL: NCT05271006
Title: COvid-19 Pandemic and Exercise for Health Care Workers (COPE HCW) Trial: A Randomized Study Examining Physical Activities and Wellbeing.
Brief Title: COVID-19 Research: COPE Trial in Health Care Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Eli Puterman, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H21-02612
Record Dates: First submitted 2022-03-02; First posted 2022-03-08 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms; Physical Inactivity
Keywords: Exercise; Intervention; mhealth; Depression; Heatlh care workers
MeSH Terms: conditions — Depression; Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Power analysis with three different effect sizes δ: .30, .40, and .50.
  Using Optimal Design Software, to detect a small effect size δ= .30 based on a two-level (non)linear growth model (six time points; level-1 residual variability = 8.798; level-1 coefficient variability = 22.548) with Power (1 - b) = .80 and alpha = .05 for 7 time points repeated measures design, 357 participants required across the four arms. With an additional 10 recruitment sites, investigators require an additional 90 participants (for the possibility of nesting or for creation of 9 dummy variables to covary locations). With a 20% expected attrition, a total of 560 HCWs will be randomized. Investigators will be employing this conservative target for this study.
  In order to detect a small effect size δ= .40 and a 20% expected attrition, a total of 366 HCWs will be randomized.
  In order to detect a small effect size δ= .50 and a 20% expected attrition, a total of 276 HCWs will be randomized.
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI will be blind to the allocation to the groups. Person sending out emails to participants to complete surveys will be blind to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Weeks 1 - 12:
  * For the duration of the study, participant will be completing any of the physical activities customizable within the Down Dog apps. He/she will be asked to complete a minimum of four 20-minute workouts per week.
  * Every two weeks, participant will receive a survey to complete.
  Week 24:
  * At week 24 (12 weeks after their initial 12-week participation in the study), participant will receive a check-in email with the final survey to complete.
  * Investigators will also record the use of the apps at week 24.
  Interventions: Behavioral: Exercise
- Waitlist control group (No Intervention): Weeks 1 - 12:
  * For the 12 weeks of the study, participant will be asked to continue their typical, pre-study daily and weekly routine, maintaining the physical activity he/she was completing before the start of the study.
  * Every two weeks, the participant will receive a survey to complete.
  Week 24:
  • At the end of the first 12 weeks that he/she have access to the suite of apps (i.e., 24 weeks following their randomization to the waitlist control group), participant will receive a check-in email with the final survey to complete.

INTERVENTIONS:
Behavioral: Exercise — The mHealth platform to be used by the exercise group is Down Dog, which has a suite of apps for yoga, HIIT, barre, and running workouts. Down Dog has agreed to provide free memberships for one year to all participants in the study. To ensure participant de-identification on the Down Dog platform, each participant will receive a Participant ID which will be pre-registered by the study coordinator on the Down Dog platform. Randomized participants will be provided instructions for downloading the apps onto their phone or a link to the website to be used on their computer. Following randomization, participants in the exercise group will be asked to engage in physical activity (using any if the Down Dog apps), 4 days a week for 20 minutes a day for 12 weeks.
  Arms: Exercise group

SUMMARY:
The present project is designed to address the problem of elevated depression and stress among health care workers (HCWs). Investigators will test the extent to which a 12-week mobile health aerobic exercise intervention (4 days/week for 20 minutes/day) impacts HCWs reported depression. Investigators propose a 2-arm (exercise and waitlist control) parallel randomised controlled trial, with 560 underactive participants recruited from Providence Health Care. Participants will complete an online questionnaire (baseline and every 2 weeks until week 12, and again at week 24) assessing depressive symptoms (primary outcome), stress, flourishing, resilience, life satisfaction, burnout, work-family spillover, , sleep quality, workplace engagement, and absenteeism (secondary outcomes).

DETAILED DESCRIPTION:
HCWs account for the largest sector of government employees in Canada. Regulated nurses - registered nurses, nurse practitioners, licensed practical nurses, and registered psychiatric nurses - constitute the most common HCW, with over 93% of HCWs being registered nurses across Canada. The most recent National Survey of the Work and Health of Nurses reported that compared with the average working Canadian, nurses work longer shifts, more overtime, more unpaid overtime, and have more conflict at work. Nurses also report greater stress, depression, more absenteeism, higher rates of medication use, and poorer physical health than the average employed Canadian. Shift work, high job strain and low autonomy have all been linked with decreased physical and mental health among nurses. Similarly, physicians are highly stressed and at risk for burnout and disease: 92% of physicians - including family medicine, medical specialists, and surgical specialists - work in urban areas and work more than 54 hours per week, excluding on-calls. A recent National Physician Health Survey, sampling over 2500 physicians, reported high levels of emotional exhaustion (26%), overall burnout (30%), depression (34%), and suicidal ideation (9-19%). Physicians experience more than twice as much high work stress (64% compared to 27%) as the general Canadian population. The mental health conditions reported by physicians is a direct consequence of their workload, which is physically demanding and accompanied by sleep deprivation.

To investigators knowledge, there are no studies that have used a mobile application promoting exercise to reduce the depressive symptomatology, psychological distress, and physical symptoms among HCWs in a hospital or home setting. Dr. Puterman's COVID-19 Pandemic and Exercise (COPE) trial (https://www.copetrial.ca/) is the first to study the impact of a mhealth-delivered program designed for physically distanced adults at the start of the pandemic. Results indicate significant treatment effects between those randomized to the active groups (who experienced a reduction in depressive symptoms over the 6-week period) compared to waitlist control (who remained elevated in depressive symptoms). Importantly, these effects were even more apparent in the adults with pre-randomization high levels of depression. Also, the group that was given access to both the HIIT and yoga apps had the highest adherence rates for trial completion (58%) compared to those who received access to either but not both apps (53% or 40% for yoga and HIIT, respectively). Considering the above, the purpose of the present study is to evaluate the uptake and adherence of a 12-week mhealth physical activity (access to all the mobile "Down Dog" apps: HIIT, yoga, barre, running) intervention in physically less active HCWs, to examine whether the intervention leads to improvement in depressive symptomatology among those randomized to the intervention versus waitlist control group. Specifically, investigators aim to focus on physical activities requiring little physical space and/or equipment that are easily completed at home, in one's neighbourhood, or in a small office using the suite of mobile apps from the company "Down Dog".

The purpose of the present study is to evaluate the uptake and adherence of a 12-week mhealth physical activity (access to all the mobile "Down Dog" apps: HIIT, yoga, barre, running) intervention in physically less active HCWs, to examine whether the intervention leads to improvement in depressive symptomatology among those randomized to the intervention versus waitlist control group. Specifically, investigators aim to focus on physical activities requiring little physical space and/or equipment that are easily completed at home, in one's neighbourhood, or in a small office using the suite of mobile apps from the company "Down Dog".

The primary objectives of this project are to test a mhealth physical activity intervention, using the "Down Dog" suite of apps, in physically less active HCWs, and to test whether the intervention leads to improvement in depressive symptomatology among those who are randomized to the intervention compared to the waitlist control group. The secondary objectives of this project are to test the intervention effects on a broader suite of mental health concepts, including stress, flourishing, resilience, life satisfaction, burnout, work-family spillover, sleep quality, and absenteeism. Thirdly, investigators seek to identify barriers and facilitators to increasing levels of physical activity during the intervention, from the perspective of stakeholders such as nurses, health service administrators, and physicians, and to determine the efficacy of the intervention, using qualitative interviews and focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who currently do not meet recommendations for a physically active lifestyle, are over the age of 18 inclusive, who are not retired, work at a PHC centre, and are without risk factors for cardiovascular events are eligible for inclusion.
* To screen for the low active participants, investigators will use the L-CAT (see Section 9.5). All participants who score 1-3 will be included in the study. Those who score 4-6 will be excluded.
* They must also work at a Providence Health Care centre.

Exclusion Criteria:

* Participants must be cleared to participate in exercise. The 2021 Physical Activity Readiness Questionnaire for Everyone (PAR-Q+; Section 9.5) will be used to minimize any risk of exercise and ensure the safety of individuals (Warburton, Jamnik, Bredin, Shephard, & Gledhill, 2018). Given that exercise is a risk factor for cardiovascular events, participants must report any family history of cardiovascular disease, stroke or myocardial infarction (American College of Sports Medicine, 2018). If participants do report a family history of cardiovascular events, they must receive a note from their family physician clearing them for moderate to high intensity training. If payment is required for this clearance, participants will be reimbursed.
* In addition, as informed consent requires individuals to be at least 18 years old, participants under the age of 18 will be excluded.
* Participants who are currently retired from their work or who do not currently work at a PHC centre are ineligible to participate.
* Participants without personal smartphones or computers, and those without internet service at home will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptomology over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention).
  The 10 Item Center for Epidemiologic Studies Depression Scale (CES-D) will be used in the baseline survey, and will be in each biweekly survey to track changes in the CES-D over the study period. The possible range in scores is 0 to 30 depending on number of symptoms, with those symptoms weighted by frequency experienced in a week. Higher scores indicating more or more frequent symptoms.

SECONDARY OUTCOMES:
Changes in psychological stress as measured by the SCSQ over the course of the exercise intervention. | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention).
  The 1 Item Statistics Canada Stress Question (SCSQ) will be used in the baseline survey and in each biweekly survey to track changes in psychological stress over the study period. The SCSQ is a 1-item question with a possible scoring of 1 (Not at all stressful) to 5 (Extremely stressful).
Changes in flourishing over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  Diener's Flourishing scale will be used in the baseline survey, and will be in each biweekly survey to track changes in flourishing over the study period. There are 8 items, phrased in a positive direction. Scores can range from 8 (strong disagreement with all items) to 56 (strong agreement with all items), with higher scores indicating individuals who have a more positive view of themselves in important areas of functioning.
Changes in life satisfaction over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  5-item Satisfaction with life scale will be used in the baseline survey, and will be in each biweekly survey to track changes in life satisfaction.
Changes in burnout as measured by the MBI-GU over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  The 16-item Maslach Burnout Inventory - General Use (MBI-GU) will be used in the baseline survey, and will be in each biweekly survey to track changes in burnout over the study period.
  The scales of the MBI-GS provide a three-dimensional perspective on burnout. In a manner similar to the MBI-HSS, a high degree of burnout is reflected in high scores on Exhaustion and Cynicism and low scores on Professional Efficacy.
Changes in resilience as measured by the BRS over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  The Brief Resilience Scale (BRS) will be used in the baseline survey, and will be in each biweekly survey to track changes in resilience over the study period. The BRS uses a mean scoring system with a possible range in scores from 1-5, higher scores indicate the individual perceives they have a better ability to 'bounce back' and recover from stressful events and/or situations.
Change in work-family spillover over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  6-item work family experience scale will be used in the baseline survey, and will be in each biweekly survey to track changes in work-family spillover over the study period.
Change in absenteeism over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  Number of days of sick leave will be asked in the baseline survey, and will be in each biweekly survey to track changes over the study period.
Change in sleep quality over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  1-item Pittsburgh Sleep Quality Index will be asked in the baseline survey, and will be in each biweekly survey to track sleep quality changes over the study period.
Changes in leisure time physical activity over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  The investigators are tracking leisure time physical activity at baseline, and biweekly (outside of the exercise intervention) using a version of the leisure score index (LSI) that was modified from the original LSI that was part of Godin's Leisure Time Exercise Questionnaire (GLTEQ). This question allows participants to tell us the frequency per week and time per exercise session of any mild, moderate, or strenuous exercise the participants have completed.
Changes in physical health symptomology over the course of the exercise intervention | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  A Physical Health item will be used in the baseline and weekly surveys to track changes in physical health (e.g. headache, backache, fever, sore throat, fatigue etc.) over the course of the study period. There are 13 physical symptoms, with the scoring based on how many symptoms were experienced in the past week. The scoring range is 0-13, with higher numbers indicating experiencing more negative physical health symptoms.
Tracking the amount of exercise variety | Tracked biweekly for 12 weeks (baseline, followed by 12 weeks of exercise intervention)
  Using the Perceived Variety in Exercise (PVE) questionnaire, the investigators are tracking how varied participants feel their exercise activities are. There are 5 items asking about exercise variety, scored 1 (false) to 6 (true), with a possible score of 5-30; higher scores indicate greater perceived variety.
Changes in use of apps over the course of the exercise intervention | Tracked weekly for 12 weeks
  Examination of adherence rate for completing 4 session of 20 minutes per week using one of the apps (running, barre, yoga, HIIT).

CONTACTS AND LOCATIONS:
Overall Officials: Eli Puterman, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification upon request and cleared for approval by principal investigator.
  All of the protocols, statistical analysis plan, informed consent form, analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4 months following trial's end, materials will be made available. following publication, all data will be made available.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for the purpose for the purpose of meta-analyses and to achieve aims in the approved proposal. Investigators of the study need to approve the proposals. Proposals should be directed to eli.puterman@ubc.ca.
URL: https://osf.io/8qfxh/

REFERENCES:
- [Background] Embriaco N, Papazian L, Kentish-Barnes N, Pochard F, Azoulay E. Burnout syndrome among critical care healthcare workers. Curr Opin Crit Care. 2007 Oct;13(5):482-8. doi: 10.1097/MCC.0b013e3282efd28a. PMID 17762223
- [Background] Martin M. Physician Well-Being: Physician Burnout. FP Essent. 2018 Aug;471:11-15. PMID 30107104
- [Background] Marjanovic Z, Greenglass ER, Coffey S. The relevance of psychosocial variables and working conditions in predicting nurses' coping strategies during the SARS crisis: an online questionnaire survey. Int J Nurs Stud. 2007 Aug;44(6):991-8. doi: 10.1016/j.ijnurstu.2006.02.012. Epub 2006 Apr 17. PMID 16618485
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Wu PE, Styra R, Gold WL. Mitigating the psychological effects of COVID-19 on health care workers. CMAJ. 2020 Apr 27;192(17):E459-E460. doi: 10.1503/cmaj.200519. Epub 2020 Apr 15. No abstract available. PMID 32295761
- [Background] Pospos S, Young IT, Downs N, Iglewicz A, Depp C, Chen JY, Newton I, Lee K, Light GA, Zisook S. Web-Based Tools and Mobile Applications To Mitigate Burnout, Depression, and Suicidality Among Healthcare Students and Professionals: a Systematic Review. Acad Psychiatry. 2018 Feb;42(1):109-120. doi: 10.1007/s40596-017-0868-0. Epub 2017 Dec 18. PMID 29256033
- [Background] Rathbone AL, Prescott J. The Use of Mobile Apps and SMS Messaging as Physical and Mental Health Interventions: Systematic Review. J Med Internet Res. 2017 Aug 24;19(8):e295. doi: 10.2196/jmir.7740. PMID 28838887
- [Background] Puterman E, Hives B, Mazara N, Grishin N, Webster J, Hutton S, Koehle MS, Liu Y, Beauchamp MR. COVID-19 Pandemic and Exercise (COPE) trial: a multigroup pragmatic randomised controlled trial examining effects of app-based at-home exercise programs on depressive symptoms. Br J Sports Med. 2022 May;56(10):546-552. doi: 10.1136/bjsports-2021-104379. Epub 2021 Sep 27. PMID 34580067
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cho E, Chen TY. The effects of work-family experiences on health among older workers. Psychol Aging. 2018 Nov;33(7):993-1006. doi: 10.1037/pag0000293. Epub 2018 Oct 11. PMID 30307262
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Derived] Boucher VG, Haight BL, Hives BA, Zumbo BD, Merali-Dewji A, Hutton S, Liu Y, Nguyen S, Beauchamp MR, Black AT, Puterman E. Effects of 12 Weeks of At-Home, Application-Based Exercise on Health Care Workers' Depressive Symptoms, Burnout, and Absenteeism: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Nov 1;80(11):1101-1109. doi: 10.1001/jamapsychiatry.2023.2706. PMID 37556150